CLINICAL TRIAL: NCT03698656
Title: Effect on Patient Quality of Life of Taking Into Account the Spiritual Dimension in Nurse's Care for Haematologic Cancers : a Pilot Study
Brief Title: Effect on Patient Quality of Life of Taking Into Account the Spiritual Dimension in Nurse's Care for Haematologic Cancers.
Acronym: SPIEVIE
Status: Completed | Type: Observational
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Other Study IDs: RC31/17/0332
Record Dates: First submitted 2018-10-01; First posted 2018-10-09 (Actual); Last update posted 2020-12-28 (Actual); Status verified 2020-12

CONDITIONS: Acute Leukemia; Lymphoma
Keywords: Spiritual dimension; Hematologic cancer; Acute leukemia; Lymphoma; Nurse interview; Quality of life
MeSH Terms: conditions — Lymphoma; Hematologic Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: Spiritual Interview — Three patient interviews (45 to 60 minutes) will be conducted by the study nurse at the beginning of the study and approximately 2 and 4 month later, according to the program of the medical care. Each interview will be conducted according the active listening method of Carl Rogers.

SUMMARY:
Pilot study on feasibility of taking into account spiritual dimension in nurse's care of patients with haematologic cancer

DETAILED DESCRIPTION:
Patients with acute leukaemia or lymphoma will be invited to have three interviews centered on spiritual issues on a six-eight months period.

The intervention consist on 3 intervention interviews conducted at the beginning of the study and approximatively 2 and 4 months later (according to the program of medical care). Quality of life (FACT-G) and spiritual well-being (FACIT-SP12) scales will be completed at the beginning (before the first intervention interview) and at the end of the study (approximately 2 month after the third intervention interview, i.e. 6 to 8 month after the first interview).

This pilot study will assess the proportion of patients who will accept to enter in the study and to complete it.

ELIGIBILITY:
Inclusion Criteria:

* Patients with acute leukaemia or lymphoma, in the first month of hospitalisation after primary diagnosis or firs relapse
* More than 17 years old
* French language
* Having signed informed consent

Exclusion Criteria:

* Patients requiring palliative care
* Important psychic vulnerability or severe psychiatric disorders

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with acute leukaemia or lymphoma during the first month after diagnosis or after first relapse hospitalised in Toulouse Cancer University Hospital
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2018-10-10 (Actual); Primary Completion 2020-10-01 (Actual); Study Completion 2020-10-01 (Actual)

PRIMARY OUTCOMES:
Rate of patients accepting to enter the study and to complete it on the 6 - 8 month period | 6-8 months
  Number of patients having entered the study with regards to the number of the contacted patients, and number of patients having completed the six-eight month study with regards to the patients having entered the study

SECONDARY OUTCOMES:
Rate of entire completion of quality of life scales | 6-8 months
  Rate of entire completion of functional assessment of cancer therapy - general and The Functional Assessment of Chronic Illness Therapy Spiritual Well-Being 12 items scales whose values will be used in order to determine the sample size of a further randomised controlled trial
Number of contacted patients with regards to the number of eligible hospitalized patients | 6-8 months

CONTACTS AND LOCATIONS:
Overall Officials: Valérie FLOUCAUD, IDE, Principal Investigator — University Hospital, Toulouse
Locations (1):
- University Hospital Toulouse, Toulouse, France

IPD SHARING:
Plan to Share IPD: No